CLINICAL TRIAL: NCT03825705
Title: Phase Ib Clinical Study on Safety and Efficacy of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsule in Patients With Advanced Biliary Adenocarcinoma/Hepatocellular Carcinoma
Brief Title: A Study on Safety and Efficacy of TQB2450 Injection Combined With Anlotinib Hydrochloride Capsule in Patients With Advanced Biliary Adenocarcinoma/Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-Ib-05
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-01

CONDITIONS: Advanced Biliary Adenocarcinoma/Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib + TQB2450 (Experimental): TQB2450 1200 mg IV on Day 1 of each 21-day cycle plus Anlotinib capsules given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: TQB2450 injection; Drug: Anlotinib

INTERVENTIONS:
Drug: TQB2450 injection — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.
Drug: Anlotinib — A multi-target receptor tyrosine kinase inhibitor

SUMMARY:
A single-arm, open-label clinical trial, focus on the safety and efficacy of TQB2450 injection combined with Anlotinib hydrochloride capsule in patients with advanced biliary adenocarcinoma/hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old; ECOG physical condition: 0 - 1 points; expected survival time more than 3 months; 2、Histologically or pathologically confirmed patients with unresectable or metastatic cholangiocarcinoma, including intrahepatic cholangiocarcinoma (IHCC), extrahepatic cholangiocarcinoma (EHCC) and gallbladder cancer (GBC), or advanced hepatocellular carcinoma (Barcelona hepatocellular carcinoma stage C, or unsuitable for stage B patients who failed to receive or receive local treatment); 3、Patients had at least one measurable lesion (RECIST 1.1); 4、Previous first-line chemotherapy failed in patients with adenocarcinoma of the biliary system. First-line chemotherapy failure is defined as disease progression during or after the last treatment, or intolerable side effects during treatment. (Note: a. The first-line treatment time is more than one cycle of combined chemotherapy drugs; B. Neoadjuvant or adjuvant chemotherapy is allowed in the early stage. If disease progression/recurrence occurs during neoadjuvant/adjuvant therapy or within 6 months after the end of treatment, neoadjuvant/adjuvant therapy is considered to be the first-line systemic chemotherapy failure for progressive diseases; C. Previous first-line standardized therapy does not include small molecular inhibitors of angiogenesis or monoclonal antibodies or drugs related to tumor immunity; Patients with hepatocellular carcinoma have not received systemic chemotherapy, molecular targeted drug therapy and immunotherapy; 5、Laboratory tests should be satisfied: routine blood tests: hemoglobin (Hb) > 80g/L (no blood transfusion within 14 days); absolute neutrophil count (ANC) > 1.5 *109/L; platelet (PLT) > 75 *109/L; biochemical tests: alanine aminotransferase (ALT) and glutamic oxaloacetate aminotransferase (AST) = 2.5 *ULN (liver metastasis of tumors, < 5 *ULN); serum total bilirubin (TBIL) = 2 *ULN (Gil) Patients with Bert syndrome, < 3 *ULN; serum creatinine (Cr) = 1.5 *ULN and creatinine clearance rate > 50 umol/L; coagulation function: activated partial thromboplastin time (APTT), international standardized ratio (INR), prothrombin time (PT) = 1.5 *ULN; Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) > 50%; Child-Pugh Liver Function Rating for Patients with Liver Cancer: A-B (< 8 points), (Child-Pugh Albumin Rating must be less than 2 points, i.e. more than 28g/L; Bilirubin Rating 1 point, TBIL < 2.0xULN; Ascites Rating < 2 points; Hepatic Encephalopathy < 1 point; Prothrombin Time Rating < 2 points); 6、Women should agree to use contraceptive measures (such as intrauterine device [IUD], contraceptive pill or condom) within 6 months of the study period and the end of the study period; serum or urine pregnancy tests are negative within 7 days before the study group and must be non-breastfeeding patients; men should agree to use contraceptive measures during the study period and within 6 months after the end of the study period; 7、The patients voluntarily joined the study and signed the informed consent with good compliance.

Exclusion Criteria:

1. Patients who had previously received treatment with target inhibitors of vascular endothelial growth factor R, including Anlotinib hydrochloride capsules, or other anti-PD-1/PD-L1/CTLA-4 antibodies or other immunotherapy against PD-1/PD-L1/CTLA-4 were treated; 2、Severe hypersensitivity was observed after administration of other monoclonal antibodies; 3、Within five years, the subjects had other malignant tumors (except cured basal cell carcinoma of skin, carcinoma in situ of prostate and carcinoma in situ of cervix); 4、There is any active autoimmune disease or history of autoimmune disease (e.g., autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; asthma patients who need bronchiectasis for medical intervention can not be included); but the following patients are allowed to enter the group: vitiligo without systemic treatment, psoriasis, alopecia, well-controlled I. In type 2 diabetes mellitus, hypothyroidism with normal thyroid function is treated by substitution therapy; 5、Immunosuppressive therapy with immunosuppressive agents or systemic or absorbable local hormones (dosage > 10mg/prednisone or other therapeutic hormones) is required for the purpose of immunosuppression, and is still in use for 2 weeks after the first administration; 6、Those with multiple factors affecting oral medication, such as inability to swallow, Post-gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc; 7、Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage; 8、Regardless of the severity, patients with any physical signs or history of bleeding, patients with bleeding or bleeding events greater than or equal to CTCAE 3 within four weeks prior to the first administration, or patients with unhealed wounds, fractures, gastric and duodenal active ulcers, ulcerative colitis, or unresected tumors have active bleeding, or may be caused as determined by the researchers. Other conditions of gastrointestinal bleeding and perforation;9、Brain metastases were detected by CT or MRI at screening, and there was a history of organ transplantation;10、Within four weeks before the start of the study, the patients received approved or in-progress antineoplastic therapy, including but not limited to chemotherapy, surgery, radiotherapy, biological targeted therapy, interventional therapy, immunotherapy and antineoplastic traditional Chinese medicine treatment (based on indications of Chinese medicine instructions, such as 2-week elution period can also be included in the group), etc. (Note: Oral targeting drugs with less than 5 half-lives or oral fluorouracil; Patients with pyridine drugs for less than 14 days, mitomycin C and nitrosourea for less than 6 weeks, and patients whose adverse events (except hair loss) caused by previous treatment did not recover to < CTCAE 1 degree;11、Patients with any serious and/or uncontrollable disease, including:(a) Patients with unsatisfactory blood pressure control (systolic blood pressure (> 150 mmHg), diastolic blood pressure (> 90 mmHg);(b) Thrombotic events, ischemic attacks, myocardial infarction, grade 2 congestive heart failure or arrhythmias requiring treatment (including QTc (> 480ms) occurred within 6 months of first administration;(C) Severe active or uncontrolled infections (> CTC AE 2 infection), tuberculosis patients;(D) Known clinical history of liver diseases, including viral hepatitis, known carriers of hepatitis B virus (HBV) must exclude active HBV infection, that is, HBV DNA positive (> 1 *104 copies/mL or > 2000 IU/mL); known hepatitis C virus infection (HCV) and HCV RNA positive (> 1 *103 copies/mL), or other decompensated hepatitis and chronic hepatitis, which require antiviral treatment. Therapy;(E) HIV positive;(F) poor control of diabetes mellitus (fasting blood sugar (> CTCAE 2);(G) Urinary routine indicated that urinary protein (++) and confirmed 24-hour urinary protein quantification (>1.0 g);12、Vaccinated with vaccines or attenuated vaccines within 4 weeks after first administration; 13、According to the judgement of the researchers, there are other factors that may lead to the termination of the study. For example, other serious diseases (including mental disorders) need to be treated together, there are serious abnormal laboratory examinations, accompanied by family or social factors, which will affect the safety of the subjects, or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate(ORR) | Up to 96 weeks
  Overall Response Rate (ORR) defined as the proportion of subjects who achieves a best response of CR or PR, assessed by RECIST1.1/irRECIST

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Gong C, Huang J, Cao D, Liu T, Cai Q, You S, Sun Y, Jiang Z, Wang W, Yang L, Zhao H, Zhang W, Zhou A. Serum BDNF helps identify favorable subgroups in HCC patients treated with PD-L1 inhibitors and anti-angiogenic TKIs. Ther Adv Med Oncol. 2025 Dec 23;17:17588359251407052. doi: 10.1177/17588359251407052. eCollection 2025. PMID 41466842
- [Derived] Zhou J, Sun Y, Zhang W, Yuan J, Peng Z, Wang W, Gong J, Yang L, Cao Y, Zhao H, Chen C, Wang W, Shen L, Zhou A. Phase Ib study of anlotinib combined with TQB2450 in pretreated advanced biliary tract cancer and biomarker analysis. Hepatology. 2023 Jan 1;77(1):65-76. doi: 10.1002/hep.32548. Epub 2022 Aug 18. PMID 35491432